CLINICAL TRIAL: NCT00215774
Title: Targeted Pharmacological Reversal of Electrical Remodeling After Cardioversion.
Brief Title: Flecainide-Short Long Study (Flec-SL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Meda Pharmaceuticals (Industry); German Research Foundation (Other)
Responsible Party: Principal Investigator, Paulus Kirchhof, Prof MD, Atrial Fibrillation Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFNET-B11
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No antiarrhythmic treatment (No Intervention): Control group
- B-Flecainide treatment (Experimental): 4 weeks treatment with flecainide
  Interventions: Drug: Flecainide
- C-Flecainide treatment (Experimental): 6 months flecainide treatment
  Interventions: Drug: Flecainide

INTERVENTIONS:
Drug: Flecainide — Flecainide 2 - 3 x 100 mg/d The main difference between the two active therapy groups is the duration of treatment.
  Other Names: Flecainide in all its approved oral preparations
  Arms: B-Flecainide treatment; C-Flecainide treatment

SUMMARY:
A randomized trial to test the hypothesis that short-term pharmacological reversal of electrical remodeling after cardioversion is equally efficient to prevent recurrent atrial fibrillation as standard long-term antiarrhythmic therapy.

DETAILED DESCRIPTION:
Details of the trial are described in a design paper published in the American Heart Journal (1).

Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia with approximately one million affected patients in Germany. Current estimates suggest that the life-time risk for AF is 30% for men and slightly less for women at the age of 40 years. Due to demographic changes in the German population, the incidence and prevalence of AF is expected to double within the next 30 years. AF almost doubles mortality and causes important morbidity, mainly due to thrombo-embolic complications and stroke. In addition, the arrhythmia in itself reduces the chronotropic adaptation of the heart to increased work load and reduces cardiac output, especially in patients with heart failure or other cardiac disease. Restoration of sinus rhythm would reduce this burden of disease.

Acute termination of AF is almost always successful by external electrical cardioversion, especially using recently optimized techniques [biphasic shock wave forms, anterior-posterior electrode position, sintered steel electrode paddles. Maintaining sinus rhythm, however, is a more difficult task. Antiarrhythmic, ion channel-blocking drugs are effective in preventing a part of recurrent episodes of AF. Their long-term use, however, is limited by pro-arrhythmic side effects which are especially apparent during long-term therapy. AF initiates major changes in atrial electrophysiology per se which have been summarized as "electrical remodeling". The main consequence of these changes is a shortening of the atrial refractory period and action potential duration. Electrical remodeling maintains AF and is related to recurrence of AF after successful cardioversion. Electrical remodeling is reversed when sinus rhythm is maintained over approximately 4 weeks after successful cardioversion. Interestingly, the vast majority of AF recurrences occur during these first few weeks after cardioversion.

Conceptually, the initial phase of "reversal" of electrical remodeling can be separated from the long-term treatment aimed at modifying the underlying substrate of AF. Classical sodium- or potassium channel blocking antiarrhythmic drugs prolong the atrial action potential even in the fibrillating atrium and may therefore support or even anticipate reversal of electrical remodeling. Such pharmacological reversal of electrical remodeling may only transiently be required, i.e. until electrical remodeling is in itself reversed by the natural restoration of normal atrial electrophysiology. Atrial action potential prolongation beyond normal values may indeed even be pro-arrhythmic. Therefore, it is tempting to treat the main electrophysiological end point of electrical remodeling, shortening of atrial action potential duration, by a limited short-term use of action potential-prolonging antiarrhythmic drugs.

Hypothesis: Targeted "pharmacological reversal" of atrial remodeling by short-term administration of action potential prolonging antiarrhythmic drugs (4 weeks therapy duration) is equally efficient and potentially safer to prevent recurrent AF after cardioversion when compared to current long-term antiarrhythmic drug therapy.

Trial design: This is a prospective, randomized, controlled, open label, parallel group multi-center investigator-initiated trial. The study medication is prescribed in an open fashion. We chose an open design in order to increase external validity ("relevance for clinical practice") of the results.

After successful cardioversion, patients will be randomized to one of three treatment groups:

Group A: No antiarrhythmic treatment

Group B: 4 weeks antiarrhythmic treatment with flecainide

Group C: Standard long term antiarrhythmic treatment (6 months) with flecainide

Group sizes were calculated to allow demonstration of non-inferiority of the two active treatment arms with a 10% boundary.

Flecainide was chosen for antiarrhythmic treatment in the Flec-SL trial because it is effective in the prevention of recurrent AF after cardioversion in the absence of major structural heart disease, has been safe as an outpatient treatment for recurrent AF, and prolongs the atrial action potential in patients with AF. In addition to its action potential-prolonging effect, flecainide induces post-repolarization refractoriness in the atria, an electrophysiological effect that may assist in the prevention of recurrent AF.

This is an investigator-initiated trial. Sponsor is the AFNET (www.kompetenznetz-vorhofflimmern.de).

Primary end point is the time to persistent AF as assessed by daily telemetric ECG recordings and confirmed by conventional Holter ECG recordings. Secondary end points include burden of AF, time to first symptomatic episode of AF, AF burden (number and duration of AF episodes), number of hospitalizations due to AF, time to termination of trial medication, number of serious adverse events including pro-arrhythmic events, and quality of life. Details of the secondary end points are indicated in the approved trial protocol.

All patients are systematically followed for 6 months by daily telemetric ECG recordings. All recordings are obtained using miniaturized ECG recorders which allow recording of a 60-second ECG and transtelephonic ECG transmission of the ECG via a toll-free number. All ECGs are received at the central analysis unit located at the Institute for Clinical Cardiovascular Research (IKKF) in Munich. Each telemetric ECG is analyzed within 24 hours of receipt at the analysis unit. The study physician is informed in case of any abnormal results within these 24 hours. Suspicion of persistent atrial fibrillation in the Tele-ECG prompts a local visit to record a Holte ECG. The Holter ECGs are centrally analyzed (blinded end point analysis). The systematic telemetric ECG monitoring allows for detection of all episodes of recurrent persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Documented persistent atrial fibrillation
* Age of 18 years
* Documented oral anticoagulation (INR ≥ 2) for at least three weeks prior to inclusion, or exclusion of left atrial thrombi by trans-esophageal echocardiography
* Written informed consent of the patient

Exclusion Criteria:

* Current therapy with antiarrhythmic agents of class I and class III other than study medication flecainide. Such antiarrhythmic treatment must be stopped five half lives prior to enrollment. Five half lives correspond to 48 hours for almost all antiarrhythmic agents. For details regarding a specific agent, this information can be obtained through the internet at www.rote-liste.de or from the Fachinformation of the specific compound.
* Long-term therapy with amiodarone within the last 6 months prior to inclusion
* Symptomatic bradycardia or symptomatic sick sinus syndrome unless treated with a permanent pacemaker
* Symptomatic higher degree AV nodal block (grade II or III) unless treated with a permanent pacemaker
* Brugada syndrome
* Typical angina pectoris symptoms at rest or during exercise
* Known untreated coronary artery disease with high-degree coronary stenosis (> 80% reduction in luminal diameter)
* Myocardial infarction within the last 3 months
* Left ventricular ejection fraction of more than 40%
* Creatinine clearance < 50 ml/min*1.73 m2 as determined by the Cockroft-Gould formula. The digital data management system will calculate this value for you during the inclusion process. For completeness of documentation, the formula is given below:
* Men: Creatinine clearance (ml/min) = (140 - age(years)) * body weight (kg) / (72 * serum creatinine level (mg/dl))
* Women: Value for men * 0,85
* Manifest hepatic insufficiency
* Hyperthyroidism or hypothyroidism manifested clinically and in laboratory tests (TSH, T3, T4)
* Females who are pregnant or breast feeding
* Females of childbearing potential who are not using a scientifically accepted method of contraception
* Participation in a clinical trial within the last 30 days. Simultaneous participation in a registry (e.g. project AB1 of the AFNET) is permitted.
* Drug addiction or chronic alcohol abuse
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical trial
* Evidence of an uncooperative attitude
* Prolongation of the QRS complex by more than 25% during flecainide treatment (measured as the difference in QRS duration between the baseline ECG and the ECG at cardioversion (34))

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2005-03; Primary Completion 2009-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
time to persistent atrial fibrillation as determined by daily telemetric ECG recordings and verified by Holter ECG recording | primary endpoint

SECONDARY OUTCOMES:
time to first symptomatic episode of AF | end of trial
AF burden (number and duration of AF episodes) | end of trial
number of hospitalizations due to AF | end of trial
time to termination of trial medication | end of trial
number of serious adverse events including pro-arrhythmic events | end of trial
quality of life | end of trial

CONTACTS AND LOCATIONS:
Overall Officials: P Kirchhof, Prof, Principal Investigator — AFNET, Kompetenznetz Vorhofflimmern; G Breithardt, Prof, Principal Investigator — AFNET, Kompetenznetz Vorhofflimmern

REFERENCES:
- [Background] Kirchhof P, Fetsch T, Hanrath P, Meinertz T, Steinbeck G, Lehmacher W, Breithardt G. Targeted pharmacological reversal of electrical remodeling after cardioversion--rationale and design of the Flecainide Short-Long (Flec-SL) trial. Am Heart J. 2005 Nov;150(5):899. doi: 10.1016/j.ahj.2005.07.020. PMID 16290956
- [Result] Kirchhof P, Andresen D, Bosch R, Borggrefe M, Meinertz T, Parade U, Ravens U, Samol A, Steinbeck G, Treszl A, Wegscheider K, Breithardt G. Short-term versus long-term antiarrhythmic drug treatment after cardioversion of atrial fibrillation (Flec-SL): a prospective, randomised, open-label, blinded endpoint assessment trial. Lancet. 2012 Jul 21;380(9838):238-46. doi: 10.1016/S0140-6736(12)60570-4. Epub 2012 Jun 18. PMID 22713626
- [Derived] Apostolakis S, Haeusler KG, Oeff M, Treszl A, Andresen D, Borggrefe M, Lip GY, Meinertz T, Parade U, Samol A, Steinbeck G, Wegscheider K, Breithardt G, Kirchhof P. Low stroke risk after elective cardioversion of atrial fibrillation: an analysis of the Flec-SL trial. Int J Cardiol. 2013 Oct 9;168(4):3977-81. doi: 10.1016/j.ijcard.2013.06.090. Epub 2013 Jul 18. PMID 23871349
- See also: Kompetenznetz Vorhofflimmern (AFNET) — http://www.kompetenznetz-vorhofflimmern.de